CLINICAL TRIAL: NCT04241809
Title: Bioaerosol Sampling of Patients With Suspected Pulmonary Tuberculosis: A Study Protocol
Brief Title: Bioaerosol Sampling in Suspected Pulmonary Tuberculosis
Status: Completed | Type: Observational
Sponsor: Desmond Tutu HIV Foundation (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Cape Town (Other); Zeteo Tech Incorporated (Unknown)
Responsible Party: Sponsor
Other Study IDs: R01AI147347-01 (NIH)
Record Dates: First submitted 2019-11-27; First posted 2020-01-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Pulmonary Tuberculosis Confirmation by Sputum Microscopy With or Without Culture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Mtb lipid and genomic containing respiratory bioaerosol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A: Notified TB with sputum laboratory confirmation: Bioaerosol Sampling: (1) direct sampling of a specific respiratory manoeuvre; and (2) indirect, following passive respiratory activity and environmental sampling.
  Repeat bioaerosol sampling will be conducted at 14 days.
  Interventions: Diagnostic Test: Bioaerosol Sampling
- B: Notified TB without sputum laboratory confirmation: Bioaerosol Sampling: (1) direct sampling of a specific respiratory manoeuvre; and (2) indirect, following passive respiratory activity and environmental sampling.
  Repeat bioaerosol sampling will be conducted at 14 days.
  Interventions: Diagnostic Test: Bioaerosol Sampling
- C: Not Notified for TB: Bioaerosol Sampling: (1) direct sampling of a specific respiratory manoeuvre; and (2) indirect, following passive respiratory activity and environmental sampling.
  Repeat bioaerosol sampling will be conducted at 14 days.
  Interventions: Diagnostic Test: Bioaerosol Sampling

INTERVENTIONS:
Diagnostic Test: Bioaerosol Sampling — Cyclone collection of exhaled bioaerosol

SUMMARY:
Tuberculosis (TB) is transmitted in bioaerosols containing Mycobacterium tuberculosis (Mtb). Mtb-containing bioaerosols are likely related to host infectiousness and central to ongoing TB transmission. No routine diagnostic assay exists to measure Mtb in bioaerosols. Furthermore, published studies of Mtb in bioaerosol samples, have been limited to individuals with sputum-positive pulmonary TB. Currently TB diagnosis is based on clinical symptoms and sputum laboratory findings. However, approximately half of all patients commencing TB treatment are sputum negative resulting in a high proportion of presumptive treatments. We therefore propose to use a sensitive sampling protocol to investigate the prevalence of Mtb-containing bioaerosols in both sputum-positive and sputum-negative TB suspects.

DETAILED DESCRIPTION:
Our pragmatic, parallel-group design is aimed at identifying viable Mtb in bioaerosols produced by individuals attending a TB clinic in Cape Town, South Africa. Bioaerosol sampling will be performed on all eligible individuals presenting with symptoms indicative of TB and repeated at 14 days if initially positive for viable Mtb. Participants will be classified into three distinct groups based on the National TB Control Program (NTBCP) criteria: Group A, TB notification with sputum-based laboratory confirmation; Group B, TB notification with empiric diagnosis; and Group C, individuals not notified. Group C individuals with detectable Mtb bioaerosol will be monitored until resolution of clinical and laboratory status. Collection of bioaerosol specimens will be via two consecutive sampling modalities: (1) direct sampling of a specific respiratory manoeuvre; and (2) indirect sampling following passive respiratory activity and environmental sampling. microscopy. Mtb genomes and mycobacterial and host lipids will be detected using droplet digital PCR and mass spectrometry analyses, respectively. The primary objective is to determine the prevalence of Mtb bioaerosols in all TB clinic attendees and in each of the mutually exclusive groups A, B and C. Secondary objectives are to investigate differences in prevalence of Mtb bioaerosol by HIV status, current isoniazid preventive therapy (IPT) use and pre and post initiation of anti-TB chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* age over 13 years
* person with suspected TB
* provision of written, informed consent (parental consent and patient assent for those aged under 18yrs)

Ages: 13 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with respiratory and/or constitutional symptoms suggestive of pulmonary TB who self-present to two TB clinics in high density peri-urban settlements in Cape Town, South Africa will be offered recruitment to the study
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Primary Aim | 12 months
  The difference in prevalence proportions of Mtb-containing bioaerosol in sputum positive and sputum negative pulmonary TB cases (Groups A & B)

SECONDARY OUTCOMES:
Secondary Aim (1) | 12 months
  The difference in numbers of viable MTB organisms in bioaerosols per liter of air sampled and per nano-liter of bioaerosol particulate volume collected in both sputum positive and sputum negative pulmonary TB cases (Groups A & B).

OTHER OUTCOMES:
Exploratory Aim (1) | 12 months
  The prevalence of MTB containing bioaerosols in TB suspects not diagnosed with clinical TB (Group C)
Exploratory Aim (2) | 12 months
  The difference in prevalence and numbers of viable MTB in subjects receiving and not receiving IPT prophylaxis.
Exploratory Aim (3) | 12 months
  The difference in prevalence and numbers of viable MTB in subjects with and without HIV-infection.
Exploratory Aim (4) | 12 months
  The difference in prevalence and numbers of viable MTB in subjects before and after TB therapy.
Exploratory Aim (5) | 12 months
  The difference in numbers of viable MTB in bioaerosol collected by direct and indirect sampling.
Exploratory Aim (6) | 12 months
  The ratio of MTB genomes (ddPCR) to viable MTB organisms (DMN-tre-positive) in MTB containing bioaerosol
Exploratory Aim (7) | 12 months
  Which MTB lipids are present in MTB containing bioaerosol

CONTACTS AND LOCATIONS:
Locations (1):
- Aerobiology Research Centre, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
The outcomes of the analysis in addition to the unprocessed data will be submitted for publication in open-source peer-reviewed journals and presented at international conferences.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Patterson B, Koch A, Gessner S, Dinkele R, Gqada M, Bryden W, Cobelens F, Little F, Warner DF, Wood R. Bioaerosol sampling of patients with suspected pulmonary tuberculosis: a study protocol. BMC Infect Dis. 2020 Aug 8;20(1):587. doi: 10.1186/s12879-020-05278-y. PMID 32770954